CLINICAL TRIAL: NCT03228927
Title: Characterization of the Facial and Gut Microbiome in Identical and Fraternal Twins With Rosacea; Comparison to Healthy Controls
Brief Title: Characterization of the Facial and Gut Microbiome in Rosacea
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: The Acne Cure Alliance (Other)
Responsible Party: Principal Investigator, Hilary Baldwin, Medical Director, The Acne Cure Alliance
Other Study IDs: 713
Record Dates: First submitted 2017-07-18; First posted 2017-07-25 (Actual); Last update posted 2017-07-26 (Actual); Status verified 2017-07

CONDITIONS: Rosacea
MeSH Terms: conditions — Rosacea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — skin swab and fecal sample
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- twin A: Sampling of the facial and fecal microbiome
  Interventions: Other: comparison of twin A to twin B
- twin B: Sampling of the facial and fecal microbiome
  Interventions: Other: comparison of twin A to twin B

INTERVENTIONS:
Other: comparison of twin A to twin B — Comparison of Twin A to Twin B

SUMMARY:
Questionnaires will be completed by each member of the twin set. A board-certified dermatologist will examine each member to categorize the type and severity of their rosacea. The facial and gut microbiome will be sampled and sent for microbial analysis.

DETAILED DESCRIPTION:
1. Twin set subjects will be administered a questionnaire regarding demographics (age, gender, state of residence, time lived together, birth order), rosacea duration, prior rosacea treatment, diet (and similarity of diet to twin), co-morbidities, signs and symptoms suggestive of cardiovascular or gastrointestinal disease/disorder.
2. Subjects will be examined by a board-certified dermatologist and global assessment, inflammatory counts and clinician's erythema score will be performed. Eyes will be examined for signs of ocular rosacea.
3. Facial microbiome sampling will be performed on-site utilizing a kit manufactured by UBiome. The skin with active rosacea will be swabbed and the swab immediately placed in sample medium. The tube is then shipped to the manufacturer for 16s rRNA shotgun metagenomics to identify resident bacterial genera and species. (16) This can be compared to their extensive library of normal controls, to the other member of the twin set and to acne subjects.
4. Subjects will be given a fecal microbiome kit for home sampling. Feces obtained from toilet paper is collected and placed in the sample medium. Subjects can either ship directly or return to the study site for shipping.

ELIGIBILITY:
Inclusion Criteria:

1. Presenting with monozygotic or dizygotic twin
2. One or both twins with facial rosacea
3. Willingness to allow facial and fecal samples to be analyzed -

Exclusion Criteria:

1. Non-twin siblings
2. Absence of facial rosacea in both twins -

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Attendees at the Twins Days Festival Monozygotic or dizygotic twin sets Facial Rosacea
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2017-08-05 (Estimated); Primary Completion 2017-08-06 (Estimated); Study Completion 2017-08-06 (Estimated)

PRIMARY OUTCOMES:
Characterization of the facial and fecal microbiome of monozygotic or dizygotic twins with facial rosacea | Single sampling of facial microbiome done on site over a 2-day Festival August 5 and 6, 2017.
  Characterization of the facial and fecal microbiome in monozygotic or dizygotic twins concordant or discordant for rosacea compared to a) each other, b) microbiome library of age-matched controls

IPD SHARING:
Plan to Share IPD: No
There is no plan to share any IPD with other researchers